CLINICAL TRIAL: NCT04715724
Title: Evaluation and Comparison of Baby Dolls for Teaching Newborn Positioning and Attachment in a Clinical Lactation Telesimulation
Brief Title: Comparison of Baby Dolls for Teaching Newborn Positioning and Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LiquidGoldConcept (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 21-001
Record Dates: First submitted 2021-01-05; First posted 2021-01-20 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Breastfeeding; Patient Simulation; High Fidelity Simulation Training
MeSH Terms: conditions — Breast Feeding | interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: All participants will evaluate the Newborn Oral Assessment and Latch Simulator (NORALSim) and one of two other baby dolls: 1) a cloth doll with a puppet-style head where the user can control the opening and closing of the mouth, and 2) a rigid, plastic doll with a static open mouth. The order of presentation of the dolls between the two back-to-back simulations and the second baby doll will be randomized.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not be aware which baby doll they will be assessing prior to presentation within the simulation. Standardized patients (SP) will know which baby doll to present during the simulations, so they will not be masked. Following the simulation, the SP will indicate which dolls were used using a blinded numbering system that will be used for data analysis by investigators and outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baby doll with remote controlled jaw (Experimental): In this arm, participants will complete a simulation using the Newborn Oral Assessment and Latch Simulator (NORALSim), which is designed to look, feel, and weigh like a healthy human newborn. The NORALSim's jaw can be remotely operated by the user to demonstrate attachment at the breast.
  Interventions: Other: Positioning and Attachment video-based simulation (telesimulation)
- Baby doll with hand controlled jaw (Active Comparator): In this arm, participants will complete a simulation using a cloth baby with a puppet-style jaw which can be opened and closed by the user to demonstrate attachment at the breast.
  Interventions: Other: Positioning and Attachment video-based simulation (telesimulation)
- Static baby doll (Active Comparator): In this arm, participants will complete a simulation using a rigid, plastic baby with a static, open mouth.
  Interventions: Other: Positioning and Attachment video-based simulation (telesimulation)

INTERVENTIONS:
Other: Positioning and Attachment video-based simulation (telesimulation) — Participants will teach a standardized patient actor (SP) to position and attach the baby doll at the breast of the Lactation Simulation Model in a video-based simulation (telesimulation)

SUMMARY:
In this baby doll comparison study, clinical lactation specialists will complete two back-to-back video-based simulations (telesimulations) focused on newborn positioning and attachment. Study participants will interact with a standardized patient educator (SP) wearing the Lactation Simulation Model and using two baby dolls in a randomized order.

DETAILED DESCRIPTION:
Identifying signs of effective newborn positioning and attachment is an essential skill for maternal-child care providers. No study has evaluated the effectiveness of commonly used baby dolls for teaching this skill. In this comparison study, clinical lactation specialists will be randomly assigned two baby dolls to evaluate in two back-to-back video-based simulations (telesimulations) with a standardized patient wearing the LiquidGoldConcept Lactation Simulation Model. Participants will complete a novel competency assessment using 3-second video clips to show specific components of positioning and attachment and evaluating whether any correction is needed and why or why not.

ELIGIBILITY:
Inclusion Criteria:

* Received IBCLC, CLC, FABM, or similar certification in clinical lactation
* At least 2 years professional experience with breastfeeding patients
* Work with lactating patients/clients at least monthly
* Work with positioning and attachment at least weekly

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Technical Skills Confirmation | Day 1
  Participants will confirm or deny whether they were able to teach specific components of newborn positioning and attachment with the baby doll.

SECONDARY OUTCOMES:
Relative realism of baby doll | Day 1
  Participants will be asked to compare the realism of the two baby dolls used in their simulation on a 30-point checklist. Respondent will rank the two baby dolls' ability to demonstrate specific components of positioning and attachment.
Satisfaction with baby dolls | Day 1
  Participants will participate in a 10-minute semi-structured interview immediately following the simulations and discuss what worked and didn't work about each baby doll for teaching newborn positioning and attachment. Interviews will be transcribed and thematically analyzed to report participant satisfaction/dissatisfaction with the baby dolls.

CONTACTS AND LOCATIONS:
Locations (1):
- LiquidGoldConcept, Ypsilanti, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Data will be aggregated for data analysis and publication.